CLINICAL TRIAL: NCT05737147
Title: Comparison of the Accuracy and Precision of a Zero Heat Flux Thermometer (SpotOnTM) Versus Pulmonary Artery Temperature Measurement in Patients Undergoing On-pump Heart Surgery: a Prospective, Multicentre, Observational Study.
Brief Title: Comparison of the Accuracy and Precision of a Zero Heat Flux Thermometer (SpotOn) Versus Pulmonary Artery Temperature.
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Carsten Michel Pedersen, Clinical nurse specialist, Rigshospitalet, Denmark
Other Study IDs: 17025426
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Temperature Monitoring; Cardiac Surgical Procedures
Keywords: Thermometers; Thoracic surgery; Perioperative monitoring; Temperature monitoring; Anesthesia; Body temperature; Cardiac surgical procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 100 adult patients of both genders scheduled for cardiac surgery: 100 adult patients of both genders scheduled for cardiac surgery with CPB for either coronary artery bypass grafting (CABG), aortic valve replacement (AVR), mitral valve replacement (MVR) or CABG + AVR.
  Interventions: Device: Zero Heat Flux Thermometer

INTERVENTIONS:
Device: Zero Heat Flux Thermometer — Comparison of the accuracy and precision of a Zero Heat Flux Thermometer (SpotOn) Versus Pulmonary Artery Temperature Measurement
  Other Names: Pulmonary Artery Temperature

SUMMARY:
In this study, we aim to compare the core temperature measured with two noninvasive ZHF thermometers and a urinary bladder thermometer against a gold standard blood temperature measured in the pulmonary artery in patients undergoing on-pump cardiac surgery. Additionally we intend to compare the reproducibility of the ZHF measurements by using two devices simultaneously in each patient.

DETAILED DESCRIPTION:
Anesthesia will be induced with fentanyl, propofol and rocuronium and maintained with sevoflurane and fentanyl or sevoflurane and remifentanil infusion. Hypotension after induction of anesthesia will be treated primarily with phenylephrine or ephedrine and secondarily with norepinephrine infusion.

After induction of anesthesia a PAC (Edwards Lifescience, Thermodilution Paceport Catheter 931F75, 7.5F (2.5 mm) 110 cm) will be inserted in the pulmonary artery and connected to a Vigilance 2-monitor. Core temperature at the tip of the PAC will be measured every minute and displayed on the monitor. Two SpotOn™ ZHF temperature monitoring probes (3M, Model 370 Temperature Monitoring System, St. Paul, MN) will be fixed on the skin of the left and right side of the forehead above the eyebrow before induction of anesthesia. These devices also measured core temperature every minute and displayed the values on two display screens. In addition a temperature-sensing indwelling urinary catheter (CovidienTM, Mon-a-ThermTM, Foly Catheter with temperature sensor 400TM) will be placed after induction of anesthesia to allow continuous drainage of urine and continuous measurement of body temperature.

Core temperatures measured by PAC, ZHF-thermometer and bladder thermometer will be recorded with an interval of 1 minute.

In all patients the core temperature are allowed to drop until going on CPB. There will be no no external warming or infusion warming before CPB. At initiation of CPB measurements will stop because during CPB core temperatures measured with PAC does not produce an accurate estimate of core temperature.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders scheduled for cardiac surgery with CPB for either coronary artery bypass grafting (CABG), aortic valve replacement (AVR), mitral valve replacement (MVR) or CABG + AVR

Exclusion Criteria:

* Exclusion criteria if any interruption of skin on the forehead, planned direct heat application to the forehead, or previous cerebral stroke, that might affect the accuracy of the ZHF device

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients of both genders scheduled for cardiac surgery with CPB for either coronary artery bypass grafting (CABG), aortic valve replacement (AVR), mitral valve replacement (MVR) or CABG + AVR
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
ZHF temperature right side versus PAC temperature. | Perioperatively
  ZHF temperature measured on the right side of the forehead versus PAC temperature.
ZHF temperature left side versus PAC temperature. | Perioperatively
  ZHF temperature measured on the left side of the forehead versus PAC temperature.
ZHF temperature right side versus ZHF temperature left side | Perioperatively
  ZHF temperature measured on the right side of the forehead versus ZHF temperature measured on the left side of the forehead
Bladder temperature versus PAC temperature | Perioperatively
  Bladder temperature versus PAC temperature

CONTACTS AND LOCATIONS:
Overall Officials: Carsten M. Pedersen, CRNA, MScN, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided